CLINICAL TRIAL: NCT05944341
Title: Articaine Success in Pulpectomy of Primary Molars With Irreversible Pulpitis in Children Under Four Years: a Randomized Controlled Trial
Brief Title: Articaine Efficiency in Pulpectomy of Children With Irreversible Pulpitis Under the Age of Four
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmad Elheeny, Assistant Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 778
Record Dates: First submitted 2023-06-23; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Dental Pulp Diseases
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Carticaine; Epinephrine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Articaine (Experimental)
  Interventions: Drug: articaine hydrochloride 4% with epinephrine 1:100 000; Drug: Lidocaine hydrochloride 2% with epinephrine 1:100 000
- Lidocaine (Active Comparator)
  Interventions: Drug: articaine hydrochloride 4% with epinephrine 1:100 000; Drug: Lidocaine hydrochloride 2% with epinephrine 1:100 000

INTERVENTIONS:
Drug: articaine hydrochloride 4% with epinephrine 1:100 000 — Local anesthetic agent
Drug: Lidocaine hydrochloride 2% with epinephrine 1:100 000 — Local anesthetic agent

SUMMARY:
A two-tailed randomized controlled trial with two parallel arms is aimed to compare success proportions of the articaine and lidocaine groups in children with irreversible pulpitis under 4 years. The participants will be randomly assigned into two equal groups (82 children per group): the control group will receive lidocaine and the intervention group will receive the articaine local anesthesia.

The direct observation tool FLACC was considered to assess pain severity. The behavior was assessed during pulpectomy procedures using the Frankl behavior rating scale (FBRS)

ELIGIBILITY:
Inclusion Criteria:

* Healthy 36-47 month-children (ASA class I or II) weighing at least 15 kilograms
* Children should be intellectually fit, and cooperative, with no behavior or communication abnormalities
* Presence of a carious maxillary or mandibular second primary molars with signs and symptoms of irreversible pulpitis

Exclusion Criteria:

* Molars with unrestorable crowns
* Molars with necrotic pulps, pathological mobility, gingival swelling or abscess, fistulous or sinus tract, or apical periodontitis

Ages: 36 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 164 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Face, Legs, Activity, Cry, Consolability pain scale | up to 24 hours
  its scores range from None/mild pain scores 0-3 Moderate pain scores 4-6 Severe pain scores 7-10

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad Elheeny, Minya, Minya Governorate, Egypt